CLINICAL TRIAL: NCT06868251
Title: Prevalence and Pattern of Comorbid Headache in Pediatric Epilepsy Patients Attending Assiut University Children Hospital.
Brief Title: Prevalence and Pattern of Headache in Pediatric Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Somia Rasheed Abdelrasoul, resident at the pediatrics department, Assiut University
Other Study IDs: headache in pediatric epilipsy
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Headache Disorders; Epilepsy
Keywords: epilepsy; headache; pediatric epilepsy
MeSH Terms: conditions — Headache Disorders; Epilepsy; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pediatric epilepsy patients with headache: This group consists of children aged 5-18 years with diagnosed epilepsy who are mentally normal and can describe their symptoms. The study aims to estimate the prevalence and characteristics of headache in these patients. Participants will undergo a comprehensive evaluation including medical history, physical and neurological examinations, and investigations such as EEG and neuroimaging. The research will assess various aspects of headache in relation to epilepsy, including onset, location, intensity, duration, and relationship to seizures, to better understand the comorbidity between headache and epilepsy in pediatric patients.

SUMMARY:
This study aims to determine the prevalence and characteristics of headaches in children with epilepsy, aged 5-18 years. Approximately 60 children will participate at Assiut University Children's Hospital. The research will involve medical history collection, physical and neurological exams, EEG review, and blood tests. The study seeks to improve understanding of the relationship between epilepsy and headaches in children, potentially leading to better treatment strategies. Participation is voluntary, and the risks are minimal.

DETAILED DESCRIPTION:
The primary aim of this observational cross-sectional study is to estimate the prevalence and characterize headaches in pediatric epilepsy patients. Secondary objectives include identifying potential risk factors and triggers associated with headaches in this population and assessing their impact on quality of life.

Participant Criteria

Inclusion criteria:

Children aged 5-18 years with epilepsy

Mentally normal and able to describe symptoms

Willing to participate in the study

Exclusion criteria:

Children unable to express symptoms due to mental retardation, psychiatric illness, or verbal disability

Children or parents who refuse to participate

Methodology Sample Size: 60 patients, calculated using Epi-info version 7 software, based on a previous study showing 45.7% headache prevalence in pediatric epilepsy patients.

Data Collection:

Detailed medical history, including neurological, cardiovascular, gastrointestinal, endocrine, and musculoskeletal aspects

Comprehensive headache history (onset, location, intensity, quality, duration, frequency, associated symptoms)

Epilepsy history (age of onset, duration, type, medication, seizure control)

General physical examination

Neurological examination

Investigations:

Electroencephalogram (EEG) using Nihon Kohden model 1200

Neuroimaging studies (MRI, CT) if available

Complete Blood Count (CBC)

ELIGIBILITY:
Inclusion Criteria:

- pediatric epilepsy patients (5:18 years of age) who are mentally normal and can describe their symptoms.

2/ Acceptance to participate in this study.

Exclusion Criteria:

- / Children who can't express their symptoms properly because of mental retardation, psychiatric illness or verbal disability.

2/ Children or Parents who refused to participate in this study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric epilepsy patients (5:18 years of age) who are mentally normal and can describe their symptoms and have epilepsy
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
headache prevelance | 1 month
  To estimate the prevalence and characters of headache in pediatric epileptic patients

IPD SHARING:
Plan to Share IPD: No